CLINICAL TRIAL: NCT04278781
Title: Phase II Study of AG-120 in IDH1 Mutant Chondrosarcoma
Brief Title: AG-120 in People With IDH1 Mutant Chondrosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-393
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Chondrosarcoma; Chondrosarcoma, Grade 2; Chondrosarcoma, Grade 3; IDH1 Gene Mutation
Keywords: Chondrosarcoma; Chondrosarcoma, Grade 2; Chondrosarcoma, Grade 3; IDH1 Gene Mutation; IDH1 Mutant Chondrosarcoma; AG-120; locally advanced chondrosarcoma; metastatic chondrosarcoma; Memorial Sloan Kettering Cancer Center; 19-393
MeSH Terms: conditions — Chondrosarcoma; Lymphoma, Follicular | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chondrosarcoma (Experimental): Participants will have locally advanced/metastatic or recurrent operable chondrosarcoma
  Interventions: Drug: AG-120

INTERVENTIONS:
Drug: AG-120 — AG-120 500 mg orally once daily days 1-28 of a 28-day cycle

SUMMARY:
This study is being done to see whether AG-120 is an effective and safe treatment for people with advanced/metastatic or recurrent chondrosarcoma that has IDH1 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Be >/= 18 years of age
* Have a histological diagnosis (fresh or archived tumor biopsy sample) of locally advanced/metastatic or recurrent operable chondrosarcoma (conventional grade 2 or 3 only) confirmed by central pathology review

  * Patients with low grade (grade 1) and dedifferentiated chondrosarcoma are ineligible
  * Patients with biopsy proven low grade (grade 1) pelvic chondrosarcoma are ineligible unless they have radiological imaging consistent with higher grade disease in which case they will be deemed potentially eligible. In such cases the pre-treatment biopsy should be taken where feasible from the area of presumed higher-grade disease to confirm grade 2 or 3 disease to confirm eligibility
  * Patients without confirmation of grade 2 or 3 disease will not be eligible for the study unless in the case where radiology features are consistent with high grade disease but a biopsy confirmation of this is not technically feasible. Such cases should be discussed with the principal investigator before enrollment onto the study
* Have a documented IDH1 gene mutation (from a fresh tumor biopsy or from archived tumor tissue) confirmed by a CLIA approved laboratory.
* Have an ECOG OS score of 0 to 2.
* Have expected survival of >/= 4 months.
* Have at least one measurable lesion as defined by RECIST 1.1, subjected who have received prior local therapy are eligible provided the measurable disease falls outside of the treatment field or within the field and has shown >/=20% growth in size since post-treatment assessment.
* Have documented radiographic disease progression within the preceding 4 months before study entry (date ICF signed).

Have recovered from toxicities associated with prior anti-cancer therapy to baseline unless stabilized under medical management (see washout time from different therapies in Exclusion Criteria section).

* Have adequate bone marrow functions as evidenced by:

  * Absolute neutrophil count >/=1,500/mm^3 or 100 x 10^9/L.
  * Hemoglobin >/=8/dL.
  * Platelets >/=100,000/mm^3 or 100 x 10^9/L.
* Have adequate hepatic function as evidenced by:

  * Serum total bilirubin </=2 x upper limit of normal (ULN), unless considered due to Gilbert's disease.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </=5 x ULN.
* Have adequate renal function as evidenced by:

  * Serum creatinine <1.5 x ULN OR
  * creatinine clearance >/= 50ml/min based on the cockcroft-gault glomerular filtration rate (GFR) estimation:
  * (140 Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
* Be able to understand and willing to sign the informed consent form and to comply with scheduled visits, treatment plans, procedures and laboratory tests, including serial peripheral blood sampling and urine sampling, during the study. A legally authorized representative may consent on behalf of a subject who is otherwise unable to provide informed consent if acceptable to and approved by the site's Institutional Review Board (IRB)
* Be able to swallow oral medication.
* Female subjects with reproductive potential must have a negative serum or urine pregnancy test prior to the start of therapy, or a confirmation from an obstetrician in case of equivocal serum pregnancy results. Females of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated) for at least 24 consecutive months (i.e., have not had menses at any time in the preceding 24 consecutive months). Women of reproductive potential, as well as fertile men and their partners who are female with reproductive potential, must agree to use 2 effective forms of contraception (including at least 1 barrier form) from the time of giving informed consent throughout the study and for 90 days (both females and males) following the last dose of study drug. Effective forms of contraception are defined as hormonal oral contraceptive, injectables, patches, intrauterine devices, intrauterine hormone-releasing systems bilateral tubal ligation, condoms with spermicide, or male partner sterilization.

Exclusion Criteria:

* Received a prior IDH1 inhibitor.
* Received systemic anticancer therapy or an investigational agent < 3 week prior to the Day 1 (washout from prior immune based anticancer therapy is 4 weeks).
* Received radiotherapy or other local intervention to metastatic sites of disease <2 weeks prior to Day 1.
* Underwent major surgery within 4 weeks of Day 1 or have not recovered from clinically significant post-surgery toxicities.
* Have known symptomatic brain metastasis requiring steroids. Subject with previously diagnosed brain metastases are eligible if they completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and have a radiographically stable disease for a least 3 months prior to study entry.

  *Note: up to 10mg per day of prednisolone or equivalent will be allowed,
* Has another concurrent active cancer requiring therapeutic intervention.
* Are pregnant or breastfeeding.
* Are taking known strong CYP3A4 inducers or sensitive CYP3A4 substrate medications with a narrow therapeutic window unless they can be transferred to other medication within >/=5 half-lives prior to dosing
* Are taking p-glycoprotein (P-gp) transporter-sensitive substrate medications with a narrow therapeutic window, unless they can be transferred to other medications within >/= half-lives prior to dosing, or unless the medications can be properly monitored during the study.
* Have an active infection requiring systemic anti-infective therapy or with an unexplained fever > 38.5 degrees C within 7 days of Day 1 (at the discretion of the investigator, subjects with tumor fever may be enrolled).
* Have any known hypersensitivity to any components of AG-120.
* Have significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association Class II or IV congestive heart failure: myocardial infraction: unstable angina; and/or stroke.
* Have LVEP <40% by ECHO and/or MUGA scan obtained within 28 days prior to the start of the study treatment.
* Have a heart-rate corrected QT interval [using Frederica's Formula] (QTcF) >/=450msec or other factor that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Bundle branch block and prolonged QTcF interval are permitted with approval of the principal investigator.
* Are taking medications known to prolong the QT interval, unless they can have transferred to other medications within >/= half-lives prior to dosing, or unless the medications can be properly monitored during the study (If equivalent medication is not available, QTcF should be closely monitored).
* Have known active hepatitis B (HBV) or hepatitis C (HCV) infections, known positive human immunodeficiency virus (HIV) antibody results, or acquired immunodeficiency syndrome (AIDS) related illness. Subjects with a sustained viral response to HCV or immunity to prior HBV infection will be permitted. Subjects with chronic HBV that is adequately suppressed per institutional practice will be permitted.
* Have any other acute or chronic medical or psychiatric condition, including recent or active suicidal ideation or behavior, or a laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Have known active inflammatory gastrointestinal disease, previous gastric resection, or lap band dysphagia, short bowel syndrome, gastroparesis or other conditions that limit ingestion or gastrointestinal absorption of drugs administered orally.
* Has a known medical history of progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 16 weeks
  Progression free survival includes both disease progression (as defined by RECIST 1.1) and death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ciara M Kelly, MBBCh, BAO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Johns Hopkins Hospital (Data Collection Only), Baltimore, Maryland
  - Columbia University (Specimen Analysis Only), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University (Data Collection Only), Columbus, Ohio
  - MD Anderson Cancer Center (Data Collection Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Ramsey DC. CORR Insights(R): Are IDH1 R132 Mutations Associated With Poor Prognosis in Patients With Chondrosarcoma of the Bone? Clin Orthop Relat Res. 2024 Jun 1;482(6):957-959. doi: 10.1097/CORR.0000000000003019. Epub 2024 Mar 6. No abstract available. PMID 38446419
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04278781/ICF_000.pdf